CLINICAL TRIAL: NCT00487747
Title: PEGASYS® (Peginterferon Alpha-2a 40KD) in Patients With HBeAg-positive and HBeAg-negative Chronic Hepatitis B
Brief Title: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) in Patients With Chronic Hepatitis B.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20003
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (1):
- Peginterferon Alfa-2a (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms sc weekly for 48 weeks

SUMMARY:
This single arm study will assess the efficacy and safety of PEGASYS in patients with chronic hepatitis B who are either treatment-naive, or who have failed lamivudine- or interferon-treatment in the past. All patients will receive PEGASYS, 180 micrograms s.c. weekly for 48 weeks, followed by 48 weeks of treatment-free follow-up. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-70 years of age;
* chronic hepatitis B;
* Hepatitis B Virus (HBV) DNA >100,000 copies/mL.

Exclusion Criteria:

* previous antiviral or interferon-based therapy for chronic hepatitis B in past 6 months;
* evidence of decompensated liver disease;
* history or evidence of a medical condition associated with chronic liver disease other than viral hepatitis;
* coinfection with hepatitis A, C or D, or HIV.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Russia (18):
  - Chelyabinsk
  - Irkutsk
  - Kazan'
  - Krasnoyarsk
  - Moscow
  - Nizhny Novgorod
  - Novokuznetsk
  - Novosibirsk
  - Rostov-on-Don
  - Saint Petersburg
  - Samara
  - Stavropol
  - Tomsk
  - Tyumen
  - Ufa
  - Volgograd
  - Yakutsk
  - Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 centers in Russia.
Pre-assignment Details: Out of 20 participants, 18 were included in the study. (4 were Hepatitis B Early Antigen [HBeAg] positive and 14 were HBeAg-negative).
Groups:
- Peginterferon Alfa-2a: Eligible participants were administered peginterferon alfa-2a [Pegasys], 180 microgram (mcg) subcutaneous (SC) once weekly for 48 weeks and were followed for next 48 weeks.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a
Started | 18
Completed | 7
Not Completed | 11
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 9
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug were included.
Groups:
- Peginterferon Alfa-2a: Eligible participants were administered peginterferon alfa-2a, 180 microgram (mcg) subcutaneous (SC) once weekly for 48 weeks and were followed for next 48 weeks.
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Hepatitis B Early Antigen (HBeAg) positive participants [Number; unit: participants] | 4
HBeAg-negative participants [Count of Participants; unit: Participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of HBeAg Positive Participants With Hepatitis B Virus Deoxyribonucleic Acid <100,000 Copies Per mL
Description: This study included four Hepatitis B Early Antigen (HBeAg) positive participants. Participants with Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) <100,000 copies/mL were reported.
Time Frame: Week 96
Population: All participants who received at least one dose of the study drug were considered for analysis.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Number of HBeAg Negative Participants With HBV DNA < 20,000 Copies Per mL
Description: This study included 14 HBeAg negative participants. Participants with HBV DNA <20,000 copies/mL were reported.
Time Frame: Week 96
Population: All participants who received at least one dose of the study drug were considered for analysis.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 14
Participants | 3

3. Secondary Outcome: Number of HBeAg Positive Participants With HBV DNA <400 Copies Per mL, HBsAg Seroconversion, Normalization of ALT, and Sustained HBe Seroconversion
Description: Hepatitis B Surface Antigen (HBsAg) seroconversion is defined as a decrease in HBsAg to undetectable levels and a gain of detectable levels of Hepatitis B surface antibody (HBsAb). Sustained HBe seroconversion is defined as loss of HBeAg and presence of hepatitis B e-antibody (HBeAb). This study included 4 HBeAg positive participants.
Time Frame: Week 96
Population: All participants who received at least one dose of the study drug were considered for analysis.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 4
Participants
  HBV DNA <400 copies/mL | 4
  HBsAg seroconversion | 0
  ALT normalization | 4
  Sustained HBe seroconversion | 4

4. Secondary Outcome: Number of HBeAg Negative Participants With HBV DNA <400 Copies/mL, HbsAg Seroconversion and Normalization of ALT
Description: Hepatitis B Surface Antigen (HBsAg) seroconversion is defined as a decrease in HBsAg to undetectable levels and a gain of detectable levels of HBsAb. This study included 14 HBeAg negative participants.
Time Frame: Week 96
Population: All participants who received at least one dose of the study drug were considered for analysis.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 14
Participants
  HBV DNA <400 copies/mL | 3
  HBsAg seroconversion | 2
  ALT normalization | 3

5. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Any Serious Adverse Events (SAEs)
Description: All participants who received at least one dose of the study drug were analysed. Number of participants with any adverse events and any serious adverse events are reported.
Time Frame: Up to Week 96
Population: Safety population included all participants who received at least one dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 18
Participants
  Any AEs | 3
  Any SAEs | 0

6. Secondary Outcome: Mean Change in Laboratory Parameters (ALT Levels)
Description: Mean Change in Laboratory parameters (ALT levels) is reported.
Time Frame: From Screening (Day 0) to Week 96
Population: Safety population included all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 18
International units per liter (IU/L)
  ALT (Week 1) | 92.9 (73.2)
  ALT (Week 2) | 97.2 (89.9)
  ALT (Week 4) | 109.4 (133.6)
  ALT (Week 8) | 81.2 (105.4)
  ALT Week 12) | 65.1 (35.9)
  ALT (Week 18) | 53.3 (26.2)
  ALT (Week 24) | 66.2 (32.3)
  ALT (Week 32) | 55 (30.2)
  ALT (Week 40) | 46 (17.6)
  ALT (Week 48) | 38.4 (18.4)
  ALT (Week 52) | 37.1 (5.1)
  ALT (Week 60) | 40.5 (15.1)
  ALT (Week 72) | 36.9 (4.5)
  ALT (Week 96) | 32.8 (8.1)

ADVERSE EVENTS:
Time Frame: Up to Week 96
Description: Safety population included all participants who received at least one dose of the study drug.
Arm/Group | Peginterferon Alfa-2a
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 3/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a (N=18)
Neutropenia (Blood and lymphatic system disorders) | 2
Depression (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.